CLINICAL TRIAL: NCT07103876
Title: Rescuing Mobility Function Through Surgical Removal of the Parathyroid Gland
Brief Title: Parathyroidectomy and Mobility Study
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB202500602; P30AG028740 (NIH)
Record Dates: First submitted 2025-07-21; First posted 2025-08-05 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-07

CONDITIONS: Hyperparathyroidism; Parathyroid; Mobility
Keywords: Physical Function; Inflammatory Biomarkers; Parathyroidectomy; Aging; Physical activity
MeSH Terms: conditions — Hyperparathyroidism; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Blood samples will be collected for plasma biomarker analysis (e.g., myokines, osteokines, and adipokines such as IL-6, myostatin, and FGF-21), as well as for standard clinical labs including calcium, parathyroid hormone (PTH), and vitamin D.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults aged 60 and above with primary hyperparathyroidism: Participants who are undergoing a parathyroidectomy at UF health

SUMMARY:
This study evaluates whether surgical removal of the parathyroid gland (parathyroidectomy) improves physical function and mobility in older adults with primary hyperparathyroidism (PHPT). PHPT, a common endocrine disorder in older adults, is associated with reduced muscle strength, mobility, and quality of life. This prospective observational study will enroll up to 80 participants aged 60 and older undergoing parathyroidectomy at UF Health. Participants will complete physical performance tests, wear an Actigraph device to assess physical activity, and provide blood samples for biomarker analysis at pre- and post-operative time points. The goal is to characterize changes in physical function and activity following surgery and to identify biomarkers that may predict mobility improvements. Findings will help inform future larger-scale studies and could expand surgical indications for PHPT in older adults.

ELIGIBILITY:
Inclusion:

* Age ≥ 60 years;
* Biochemical diagnosis of hypercalcemic (corrected serum calcium >10.2 mg/dL or ionized serum calcium >1.31 mmol/dL or 5.2 mg/dL on at least one serum sample) primary hyperparathyroidism as determined by board-certified endocrinologist or endocrine surgeon;
* Undergoing parathyroidectomy at UF Health;
* Willing and able to give informed consent.

Exclusion:

* Failure to provide informed consent;
* Biochemical diagnosis of eucalcemic primary hyperparathyroidism (corrected serum calcium ≤10.2 mg/dL or ionized serum calcium ≤1.31 mmol/dL or 5.2 mg/dL on at least one serum sample);
* Elected not to undergo parathyroidectomy at UF Health;
* Major surgery as deemed by principal investigator or hip/knee replacement in the past 6 months;
* Fractures to the hands, arms or legs within the last 6 months;
* Traumatic accident (i.e. motor vehicle collision, fall from elevation, etc.) resulting in orthopedic trauma or requiring prolonged immobilization (>2 weeks) within the last 6 months;
* Blood transfusion within the past 3 months;
* Self-reported myocardial infarction, cerebrovascular accident, or unstable angina within the past 6 months;
* NYHA Class 3 or 4 congestive heart failure;
* Major psychiatric disorder;
* Cancer requiring treatment in the past 1 year (including metastatic cancer), except for locally treated non-melanoma skin cancers or cancers that have clearly been cured or in the opinion of the investigator carry an excellent prognosis (e.g., Stage 1 cervical cancer);
* Renal failure requiring hemodialysis or peritoneal dialysis
* Use of bone-modifying therapies (alendronate [Fosamax], zoledronic acid [Reclast], denosumab [Prolia or Xgeva], or romosozumab [Evenity]) within 1 month of planned surgery
* Planning to permanently leave the area within 3 months of parathyroidectomy;
* Vision or hearing impairment - defined as unable to read or listen/follow instructions despite the use of maximal assistive devices (i.e. contact lenses, glasses, hearing aids, etc.)
* Participating in another clinical trial or has received an investigational product within 30 days prior to screening/enrollment.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll adults aged 60 years and older with a confirmed biochemical diagnosis of hypercalcemic primary hyperparathyroidism (PHPT) who are scheduled to undergo parathyroidectomy at UF Health. Eligible participants must be able and willing to provide informed consent and complete all study procedures, including pre- and post-operative physical assessments and blood draws.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Distance Walked in Six-Minute Walk Test (6MWT) | At pre-operative assessment and at 3 month post-operative assessment
  Measures walking endurance and aerobic capacity by recording the distance walked in six minutes along a 20-meter course.
Short Physical Performance Battery Score | At pre-operative assessment and at 3 month post-operative assessment
  A composite test assessing balance, gait speed (4-meter walk), and lower body strength (chair stands). Higher scores reflect better function.
Isokinetic Knee Strength (Biodex) | At pre-operative assessment and at 3 month post-operative assessment
  Assesses lower limb muscle strength and endurance using a dynamometer. Reports peak torque and fatigue index.
Grip Strength | At pre-operative assessment and at 3 month post-operative assessment
  Handgrip strength is measured using a dynamometer as a marker of overall muscle strength and frailty risk.
Intensity of Movement using ActiGraph Accelerometry | At pre-operative assessment and at 3 month post-operative assessment
  An objective measure of free-living physical activity using a wearable hip device that captures intensity of movement over 7 days.
Frequency of Movement using ActiGraph Accelerometry | At pre-operative assessment and at 3 month post-operative assessment
  An objective measure of free-living physical activity using a wearable hip device that captures frequency of movement over 7 days.
Duration of Movement using ActiGraph Accelerometry | At pre-operative assessment and at 3 month post-operative assessment
  An objective measure of free-living physical activity using a wearable hip device that captures duration of movement over 7 days.
CHAMPS Questionnaire Score | At pre-operative assessment and at 3 month post-operative assessment
  A validated self-report tool for older adults that measures weekly frequency and duration of common physical activities.
Pasieka Parathyroidectomy Assessment of Symptoms (PAS) | At pre-operative assessment and at 3 month post-operative assessment
  A validated 13-item questionnaire measuring severity of neurocognitive and neuromuscular symptoms common in PHPT, such as fatigue, irritability, and memory loss.
Concentration of Plasma Cytokine Biomarkers | Blood work will be collected at the pre-operative assessment, the 2 week post-operative assessment, 3 month post-operative assessment and the 6 month post-operative assessment
  Blood-based analysis of myokines (e.g., IL-6, myostatin, LIF, irisin), osteokines (e.g., IGF-1, FGF-21, osteocalcin), and adipokines (e.g., adiponectin, TNF-α) associated with muscle-organ crosstalk, inflammation, and mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical and Translational Research Building, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided